CLINICAL TRIAL: NCT06716580
Title: EQUAL: EGFR ctDNA QUantative Assessment for Lung Cancer Screening in Asian and Latinx Populations
Acronym: EQUAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Boston Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Narjust Florez, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-415
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; EGFR Gene Mutation
Keywords: Lung Cancer; EGFR Gene Mutation; EGFR-related lung cancer; EGFR positive lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Biological Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ctDNA Assay (Experimental): All participants will be asked to provide blood samples and are administered a baseline questionnaire. The blood sample will be tested using the investigational ctDNA assay. If the investigational test is positive, these participants will be followed up by CLIA verification of results. A positive CLIA result will be followed up by a lung CT scan. A positive CT scan will be followed up by referral for further evaluation. A negative CT scan will be followed up by a repeat scan in 12 months. Participants will be notified of results.
  Additionally, participants may participant in optional studies: 1) One-time survey regarding perception of lung cancer screening and ctDNA testing, 2) Virtual focus group, 3) Blood banking study
  Interventions: Device: Circulating Tumor DNA (ctDNA) Assay

INTERVENTIONS:
Device: Circulating Tumor DNA (ctDNA) Assay — Screening investigational blood test to test for EGFR L858R and exon 19 deletions, which comprise 85-90% of total EGFR mutations. A positive or indeterminate investigational test will be followed up by CLIA verification of results. A positive or indeterminate CLIA result will be followed up by a lung CT scan. A positive CT scan will be followed up by referral for further evaluation. A negative CT scan will be followed up by a repeat scan in 12 months.

SUMMARY:
This research study is studying a new blood test to screen for Epidermal Growth Factor Receptor (EGFR) positive lung cancer in healthy individuals at risk for the disease and who cannot undergo regular lung cancer screening.

The name of the test used in this research study is:

-Circulating free DNA (cfDNA) Assay

DETAILED DESCRIPTION:
The goal of this research study is to evaluate the feasibility of a novel EGFR blood plasma ctDNA screening test among East Asian and Latinx participants at risk for lung cancer and ineligible for regular lung cancer screening. The test looks for a gene change called Epidermal Growth Factor Receptor (EGFR), specifically EGFR L858R and exon 19 deletions, which comprise 85-90% of total EGFR mutations. This study seeks to determine if it is possible to use the blood test to detect this type of lung cancer that might not yet show symptoms.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, and an optional questionnaire and/or focus group.

It is expected that about 1000 people will participate in the blood sample collection, 100 individuals in the survey, and 20 individuals in the focus groups.

ELIGIBILITY:
Inclusion Criteria (Aims 1, 2, and 3) for Group 1 (50 through 80 years of age):

* Non-tobacco using (currently)
* Self-identify as East Asian (including Southeast Asian) or Hispanic/Latinx.
* East Asian includes those who self-identify as Chinese, Japanese, Korean, Taiwanese, Malaysian
* Southeast Asian includes those who self-identify as Cambodian, Thai, Vietnamese, Filipino
* Latinx includes those who self-identify as a person of Central or South American and the Caribbean including, Cuban, Puerto Rican, and Dominican culture or origin, excluding individuals originating from Spain
* Aims 1 and 2: Able to complete and understand the study's informed consent in English, Mandarin, Cantonese, Japanese, Korean, Vietnamese, Spanish, Portuguese, or Cape Verdean
* Aim 3: Able to complete and understand the study's informed consent and participate in a focus group in English, Mandarin, Vietnamese, or Spanish.

Inclusion Criteria (Aims 1, 2, and 3) for Group 2 (40 through 49 years of age):

* Non-tobacco using (currently)
* Self-identify as East Asian (including Southeast Asian) or Latinx, if any of the following criteria are met:

  * Family history of EGFR positive LC L858R or exon 19
  * Personal history of remote cancer that is not LC or other thoracic malignancies, including thymoma, thymic carcinoma, or sarcoma, as long as it was resolved over 5 years ago
  * History of TB, asthma requiring daily inhaled corticosteroids or chronic bronchitis
  * Symptoms of lung cancer for the past month, including hemoptysis, unexplained weight loss, voice hoarseness, cough or worsening cough, dyspnea or worsening dyspnea
* Excluding individuals who concurrently present with fever, covid/influenza/RSV/adenovirus infection, runny nose, sore throat, productive cough with green or yellow sputum
* Aims 1 and 2: Able to complete and understand the study's informed consent in English, Mandarin, Cantonese, Japanese, Korean, Vietnamese, Spanish, Portuguese, or Cape Verdean
* Aim 3: Able to complete and understand the study's informed consent and participate in a focus group in English, Mandarin, Vietnamese, or Spanish.

Exclusion Criteria (Aims 1, 2, and 3) for Groups 1 and 2:

* Having had a chest CT scan in the last 3 years or having an anticipated chest CT scan during the enrollment period.
* Having a current cancer or history of cancer within the last 5 years, excluding localized non-melanoma skin cancer and breast ductal carcinoma in situ.
* More than 400 lifetime cigarettes (i.e., 20 packs) of smoking or tobacco use
* Adults unable to provide informed consent
* Individuals <40 years of age
* Prisoners
* Pregnant women
* Personal diagnosis of lung cancer
* Not able to be compliant with study requirements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Non-Small Cell Lung Cancer | 2 years
  The proportion of participants with a positive assay result who are subsequently diagnosed with lung cancer through clinical pathology, among all participants tested with the assay.

SECONDARY OUTCOMES:
Testing Turnaround Time | Up to 2 years
  The duration from the time of blood draw to the release of the ctDNA testing results to the study team.
Recruitment Acceptability | Up to 2 years
  Determining proportion of screened patients who are eligible and who consent to the trial at each collaboration site
Barriers to Sample Acquisition | Up to 2 years
  Examining barriers impeding scale-up of sample collection, handling, and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Narjust Florez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Steward St. Elizabeth's, Brighton, Massachusetts
  - Dana-Farber Cancer Instiute Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Cancer Institute South Shore, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu